CLINICAL TRIAL: NCT02111330
Title: Randomized, Double Blind, Placebo Controlled, Parallel Groups Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of PBF -509 (80 mg, 160 mg and 240 mg) "After Multiple Oral Doses" in Healthy Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of PBF -509 (80 mg, 160 mg and 240 mg) "After Multiple Oral Doses" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Palo Biofarma, S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIBSP-PBF-2013-155; 2013-005035-25 (EudraCT Number)
Record Dates: First submitted 2014-03-20; First posted 2014-04-11 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson Disease
Keywords: Adenosine A2a receptor antagonist; adenosine receptor modulator; Cancer
MeSH Terms: conditions — Parkinson Disease; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Dose I - 80 mg PBF-509 (Experimental): one 80 mg PBF-509 capsule
  Interventions: Drug: PBF-509
- Dose I - Placebo (Placebo Comparator): one Placebo capsule
  Interventions: Drug: Placebo
- Dose II - 160 mg PBF-509 (Experimental): Two 80 mg PBF-509 capsule
  Interventions: Drug: PBF-509
- Dose II - Placebo (Placebo Comparator): Two Placebo capsule
  Interventions: Drug: Placebo
- Dose III - 240 mg PBF-509 (Experimental): three 80 mg PBF-509 capsule
  Interventions: Drug: PBF-509
- Dose III - Placebo (Placebo Comparator): Three Placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBF-509
  Arms: Dose I - 80 mg PBF-509; Dose II - 160 mg PBF-509; Dose III - 240 mg PBF-509
Drug: Placebo
  Arms: Dose I - Placebo; Dose II - Placebo; Dose III - Placebo

SUMMARY:
Study to assess the safety and tolerability of three doses of PBF-509 (80 mg, 160 mg and 240 mg) after repeated (8 days) single daily oral dose administration in young male and female healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females subjects, 18-45 years (inclusive) of age at the time of enrollment.
* Females must be of non-childbearing potential (i.e., surgically sterile) or have to use contraceptive measures (non-hormonal) such as condom, diaphragm or cervical/vault cap with spermicide. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom/spermicide, in addition to having their female partner use some contraceptive measures.
* Clinically acceptable blood pressure and pulse rate in supine and standing position. Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
* Body weight within normal range (Quetelet's index between 19 and 26) expressed as weight (kg) / height (m2).
* Able to understand the nature of the study and comply with all their requirements.
* Free acceptance to participate in the study by obtains signed informed consent form approved by the Ethics Committee of the Hospital (CEIC).

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* Background or clinical evidence of chronic diseases.
* Acute illness two weeks before drug administration.
* Having undergone major surgery during the previous 6 months.
* Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication
* History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 g for men or 24 gr/day for women or high consumption of stimulating beverages (> 5 coffees, teas or coca cola drinks/ day)
* Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
* Need of any prescription medication within 14 days prior to the administration of the drug and non prescription medication or herbal medicines within 7 days prior to the administration of the drug.
* Participation in other clinical trials during the previous 90 days in which an investigational drug or a commercially available drug was tested.
* Having donated blood during 4 weeks period before inclusion in the study.
* Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract.
* 12 lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥ 120 msec and QTc ≥ 440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
* Symptoms of a significant somatic or mental illness in the four week period preceding drug administration.
* History of hepatitis HBV and / or HCV and / or positive serology results which indicate the presence of hepatitis B surface antigen and / or detectable HCV ribonucleic acid (RNA).
* Positive results from the HIV serology.
* Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation.
* Positive results of the drugs at screening period or the day before starting treatment period. A minimum list of drugs that will be screened for include Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the Principal Investigator).
* Known hypersensitivity to the study drug or the composition of the galenical form.
* History of psychiatric diseases or epileptic seizures
* Females with positive results from the pregnancy test or breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | day 0-9

SECONDARY OUTCOMES:
Pharmacokinetic Profile Analysis (Plasma concentrations) | day 0-9

CONTACTS AND LOCATIONS:
Overall Officials: Juan Martínez Colomer, MD, Principal Investigator — CIM Sant Pau - I.I.B. Sant Pau
Locations (2):
- Spain (2):
  - CIM Sant Pau - I.I.B. Sant Pau, Barcelona, Barcelona
  - Palobiofarma S.L. (molecule owner), Mataró, Barcelona